CLINICAL TRIAL: NCT06533384
Title: PARPi or Capecitabine Combined With PD-1 Inhibitors Was Selected Based on the Germline BRCA1/2 Mutation vs. PD-1 Inhibitors Alone as Adjuvant Therapy in High-risk Non-pCR TNBC
Brief Title: PARPi or Capecitabine Combined With PD-1 Inhibitors as Adjuvant Therapy in High-risk TNBC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-800
Record Dates: First submitted 2024-04-06; First posted 2024-08-01 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2023-11

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental ARM (Experimental): In the experimental group, patients with confirmed deleterious mutations based on germline BRCA1/2 status receive a combination of Fuzuloparib and Camrelizumab as adjuvant therapy. Patients without germline BRCA1/2 deleterious mutations receive a combination of capecitabine and Camrelizumab as adjuvant therapy.
  Interventions: Drug: As per the germline BRCA1/2 mutation status, the selection of either Fuzuloparib or capecitabine in combination with Camrelizumab is made for adjuvant therapy.
- Control ARM (Active Comparator): 9 cycles of Camrelizumab as adjuvant therapy.
  Interventions: Drug: As per the germline BRCA1/2 mutation status, the selection of either Fuzuloparib or capecitabine in combination with Camrelizumab is made for adjuvant therapy.; Drug: 9 cycles of Camrelizumab as adjuvant therapy.

INTERVENTIONS:
Drug: As per the germline BRCA1/2 mutation status, the selection of either Fuzuloparib or capecitabine in combination with Camrelizumab is made for adjuvant therapy. — As per the germline BRCA1/2 mutation status, the selection of either Fuzuloparib or capecitabine in combination with Camrelizumab is made for adjuvant therapy.
Drug: 9 cycles of Camrelizumab as adjuvant therapy. — 9 cycles of Camrelizumab as adjuvant therapy.
  Arms: Control ARM

SUMMARY:
In TNBC patients who have completed neoadjuvant immunotherapy and local treatment, a 9-cycle regimen of PD-1 inhibitor adjuvant immunotherapy is currently considered the standard approach. Based on the classification according to their BRCA mutation status, patients with BRCA mutations choose the PD-1 inhibitor + PARPi regimen, while patients without BRCA mutations opt for the PD-1 inhibitor + capecitabine regimen. Compared to monotherapy with PD-1 inhibitors, these combination regimens may offer improved efficacy and acceptable tolerability. This study is designed as a prospective, randomized, controlled, open-label, single-center phase III trial aimed at assessing the efficacy and safety of selecting PARPi or capecitabine in combination with PD-1 inhibitors based on germline BRCA1/2 mutations as adjuvant therapy in high-risk TNBC patients who have achieved non-pCR after completion of neoadjuvant immunotherapy in conjunction with chemotherapy and local treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive breast cancer.
* Negative expression of estrogen receptor (ER) and progesterone receptor (PR) according to immunohistochemistry (i.e., tumor cells showing positive staining in less than 1% of all tumor cells).
* Negative human epidermal growth factor receptor 2 (HER2) status as determined by immunohistochemistry: HER2 score of 0/1+ or, if the score is 2+, HER2/CEP17 ratio less than 2.0 or HER2 gene copy number less than 4, as confirmed by in situ hybridization (ISH).
* Clinical tumor staging: T1c, N1-N2 or T2, N0-N2 or T3, N0-N2 or T4a-d, N0-N2.
* The subjects were required to have good organ function, as evidenced by the following tests conducted within 7 days before randomization:

Hematology examination (excluding blood transfusion or use of hematopoietic stimulating agents for correction):

* Hemoglobin (Hb) ≥ 90 g/L.
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
* Absolute lymphocyte count (ALC) ≥ 0.5 × 109/L.
* Platelet count (PLT) ≥ 100 × 109/L.
* White blood cell count (WBC) ≥ 3.0 × 109/L and ≤ 15 × 109/L.

Serum biochemistry examination (excluding recent blood transfusion or albumin administration):

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of normal (ULN).
* Alkaline phosphatase (ALP) ≤ 2.5 ULN.
* Total bilirubin (TBIL) ≤ 1.5 ULN.
* Serum creatinine (Cr) ≤ 1.5 ULN, with creatinine clearance (CrCL) ≥ 50 mL/min (calculated using the Cockcroft-Gault formula).
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 ULN, and international normalized ratio (INR) ≤ 1.5 ULN (if not receiving anticoagulant therapy).

  * Thyroid-stimulating hormone (TSH) within the normal range; if TSH is abnormal, levels of free triiodothyronine (FT3) and free thyroxine (FT4) should be examined. If FT3/FT4 results are not available, T3 and T4 measurements can be considered, and if T3/T4 levels are within the normal range, the subject can be included.
  * Urine analysis: Urinary protein < 2+; if urinary protein is ≥ 2+, a 24-hour urine protein quantification should demonstrate protein ≤ 1g.
  * Cardiac echocardiography: Left ventricular ejection fraction (LVEF) ≥ 55%.
  * 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 msec.
  * Women of childbearing potential must have a negative serum pregnancy test within 3 days prior to initiating medication, and they and their partners must agree to use highly effective methods of contraception during the study and for 180 days after the last administration of the investigational drug.
  * Voluntary participation in the clinical trial and signing of the informed consent form are required.

Exclusion Criteria:

* Known history of allergy to the components of the investigational drug.
* Previous receipt of antitumor treatment or radiation therapy for any malignancy (excluding previously cured cervical carcinoma in situ and basal cell carcinoma).
* Undergone major surgery unrelated to breast cancer within the past 4 weeks, or patients who have not fully recovered from such surgery.
* Inability to swallow, intestinal obstruction, or other factors that may affect the administration and absorption of the medication.
* Severe cardiac disease or discomfort that prevents treatment.
* Presence of mental illness or substance abuse that interferes with compliance.
* Pregnant or breastfeeding women.
* Concurrent participation in other clinical trials.
* Subjects deemed by the investigator to have conditions that pose a serious risk to the safety of the participant or may affect the completion of the study, or individuals who are considered unsuitable for inclusion based on other reasons.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 310 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
IDFS | Up to approximately 5 years
  invasive disease free survival

SECONDARY OUTCOMES:
OS | Up to approximately 5 years
  Overall survival
DDFS | Up to approximately 5 years
  Distant Disease Free Survival
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Up to approximately 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Kun Wang, MD, Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Department of Breast Cancer, Cancer Center, Guangdong Provincial People's Hospital (Guangdong Academy of Medical Sciences), Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No